CLINICAL TRIAL: NCT04569201
Title: Endoscopic and Endoscopic-Assisted Microsurgery of Intraventricular Lesions: Efficacy of Technique and Outcome Assessment
Brief Title: Endoscopic and Endoscopic-Assisted Microsurgery of Intraventricular Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nour Imam, Assistant Lecturer (Principal Investigator), Assiut University
Other Study IDs: Intraventricular Endoscopy
Record Dates: First submitted 2020-09-21; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Endoscopy in Intraventricular Lesions
MeSH Terms: interventions — Endoscopes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Procedure: Endoscope — The use of the neuro endoscope in excision of intraventricular lesions either alone or in assistance of the surgical microscope

SUMMARY:
* Assess the efficacy of the endoscope as a single tool or as an adjuvant tool to the microscope in intraventricular procedures.
* Evaluate the limitations of the endoscope in these procedures.
* Review the outcome of endoscopic and/or endoscopic assisted microsurgical intraventricular procedures.
* Achieve a verdict in the long-standing controversy about the most effective, least invasive, and optimal way to resect intraventricular lesions, can the endoscope rival the surgical microscope?

DETAILED DESCRIPTION:
Lesions within the ventricular system present a challenge to neurosurgeons (1). Their deep location and proximity to eloquent neurovascular anatomy complicate surgical approach and resection (2). Microsurgery remains the gold standard for the treatment of intraventricular tumors, but microsurgical approaches are not without limitations (3). With the use of the operative microscope, most lesions of the lateral and third ventricles are accessed by a craniotomy and either a transcortical or interhemispheric transcallosal approach. These approaches are associated with brain retraction that can result in seizures, focal neurologic deficits, and cognitive impairment (1). Also with standard microsurgical techniques, complete resection is sometimes not achieved either because of nonvisualization of hidden parts of the tumor or requirement of significant retraction of the neurovascular structures which is potentially hazardous (4). The addition of the endoscope for resection of intraventricular lesions has been described and represents a minimally invasive approach that limits brain retraction and provides direct lesion visualization (1,5,6). The recent development of endoscopic instrumentation has greatly enhanced microsurgical access to the ventricular system and would allow enhanced microsurgical access, minimize the size of the transcortical corridor, and reduce brain retraction during removal of challenging intraventricular lesions performed with the surgical microscope (7). The application of the endoscope can be used in the treatment of intraventricular lesions as arachnoid cyst with intraventricular extensions, colloid cysts, biopsies and intraventricular brain tumor removal (8). Reestablishment of CSF communication pathways is also possible endoscopically when patients develop obstructive hydrocephalus due to their intraventricular pathology (1). The biggest issues when it comes to a pure endoscopic approach concern the size and extent of the lesion, possibility of complete cure or at least long-term control of the disease, and the presence of remnants that were not completely excised (8) , However, The desire for a less invasive technique and an effective surgical approach to intraventricular pathology has directed the attention of many in the neurosurgical community towards the introduction of the endoscope as an adjuvant to or even a replacement for the microscope in intraventricular surgery (5) and consequently, neuroendoscopy has grown rapidly in the last 25 years as a therapeutic modality in the treatment of intraventricular pathologies (9,10).

ELIGIBILITY:
Inclusion Criteria:

* Intraventricular arachnoid cysts
* Intraventricular colloid cysts
* Intraventricular tumors.

Exclusion Criteria:

* Intraventricular lesions extending outside the ventricle (exception to arachnoid cysts)
* Patients who are unfit for any neurosurgical interventions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: PAtients with intraventricular lesions, presented to The Neurosurgery Department, At Assiut University Hospital in Assiut, Egypt
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Early Clinical outcome using Glasgow Outcome Scale | Early outcome: 24 hours post-operatively.
  Assessment of the post operative mortality and morbidity using:
  Glasgow Outcome Scale:
  1. Death:Self-explanatory
  2. Persistent vegetative state: Coma or severe deficit rendering the patient totally dependent
  3. Severe disability: Significant neurological deficit interfering with daily activities or prevents return to employment
  4. Moderate disability:Minor neurological deficit not interfering with daily functioning or work
  5. Good recovery:Returned to the original functional level with no deficit
Early Clinical outcome using Modified Rankin Scale | Within 6 weeks after surgery.
  The Modified Rankin Scale (mRS) is used to measure the degree of disability in patients, as follows:
  * 0: No symptoms at all
  * 1: No significant disability despite symptoms; able to carry out all usual duties and activities
  * 2: Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  * 3: Moderate disability; requiring some help, but able to walk without assistance
  * 4: Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  * 5: Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  * 6: Dead
Late outcome assessment | within 6 months after surgery
  Within six months, assessment of the performance of the patient with modified rankin scale.

REFERENCES:
- [Background] Nduom EK, Sribnick EA, Ormond DR, Hadjipanayis CG. Neuroendoscopic Resection of Intraventricular Tumors and Cysts through a Working Channel with a Variable Aspiration Tissue Resector: A Feasibility and Safety Study. Minim Invasive Surg. 2013;2013:471805. doi: 10.1155/2013/471805. Epub 2013 Jun 13. PMID 23844287
- [Background] Yasargil MG, Abdulrauf SI. Surgery of intraventricular tumors. Neurosurgery. 2008 Jun;62(6 Suppl 3):1029-40; discussion 1040-1. doi: 10.1227/01.neu.0000333768.12951.9a. PMID 18695523
- [Background] Barber SM, Rangel-Castilla L, Baskin D. Neuroendoscopic resection of intraventricular tumors: a systematic outcomes analysis. Minim Invasive Surg. 2013;2013:898753. doi: 10.1155/2013/898753. Epub 2013 Sep 26. PMID 24191196
- [Background] Singh I, Rohilla S, Kumar P, Krishana G. Combined microsurgical and endoscopic technique for removal of extensive intracranial epidermoids. Surg Neurol Int. 2018 Feb 14;9:36. doi: 10.4103/sni.sni_392_17. eCollection 2018. PMID 29527394
- [Background] Cappabianca P, Cinalli G, Gangemi M, Brunori A, Cavallo LM, de Divitiis E, Decq P, Delitala A, Di Rocco F, Frazee J, Godano U, Grotenhuis A, Longatti P, Mascari C, Nishihara T, Oi S, Rekate H, Schroeder HW, Souweidane MM, Spennato P, Tamburrini G, Teo C, Warf B, Zymberg ST. Application of neuroendoscopy to intraventricular lesions. Neurosurgery. 2008 Feb;62 Suppl 2:575-97; discussion 597-8. doi: 10.1227/01.neu.0000316262.74843.dd. PMID 18596446
- [Background] Souweidane MM, Luther N. Endoscopic resection of solid intraventricular brain tumors. J Neurosurg. 2006 Aug;105(2):271-8. doi: 10.3171/jns.2006.105.2.271. PMID 17219833
- [Background] Harris AE, Hadjipanayis CG, Lunsford LD, Lunsford AK, Kassam AB. Microsurgical removal of intraventricular lesions using endoscopic visualization and stereotactic guidance. Neurosurgery. 2005 Jan;56(1 Suppl):125-32; discussion 125-32. doi: 10.1227/01.neu.0000146227.75138.08. PMID 15799800
- [Background] Brunori A, de Falco R, Delitala A, Schaller K, Schonauer C. Tailoring Endoscopic Approach to Colloid Cysts of the Third Ventricle: A Multicenter Experience. World Neurosurg. 2018 Sep;117:e457-e464. doi: 10.1016/j.wneu.2018.06.051. Epub 2018 Jun 26. PMID 29959067
- [Background] Yadav YR, Parihar V, Sinha M, Jain N. Endoscopic treatment of the suprasellar arachnoid cyst. Neurol India. 2010 Mar-Apr;58(2):280-3. doi: 10.4103/0028-3886.63772. PMID 20508350
- [Background] Romano A, Chibbaro S, Marsella M, Oretti G, Spiriev T, Iaccarino C, Servadei F. Combined endoscopic transsphenoidal-transventricular approach for resection of a giant pituitary macroadenoma. World Neurosurg. 2010 Jul;74(1):161-4. doi: 10.1016/j.wneu.2010.02.024. PMID 21300008